CLINICAL TRIAL: NCT06374680
Title: Randomized Controlled Trial: Comparison of Radiological and Axial Pain Outcome Between C3-6 Laminoplasty and C3 Laminectomy With Cervical Laminoplasty
Brief Title: C3 Laminectomy With Cervical Laminoplasty
Status: Withdrawn | Type: Observational
Why Stopped: This is because the same research has already been done.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chun Kee Chung, professor, Seoul National University Hospital
Other Study IDs: C3 ectomy
Record Dates: First submitted 2017-08-24; First posted 2024-04-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- C3 laminectomy: laminectomy at C3 level and laminoplasty at C4-6 level
  Interventions: Procedure: laminectomy at C3 level
- C3 laminoplasty: laminoplasty at C3-6 level
  Interventions: Procedure: laminectomy at C3 level

INTERVENTIONS:
Procedure: laminectomy at C3 level — laminectomy at C3 level

SUMMARY:
1. Background In cervical stenosis, cervical laminoplasty from the third to sixth cervical vertebrae is widely used. However, the muscles attached to the C2, which play an important role in the movement of our neck, are frequently damaged during the C3 laminoplasty. In contrast, cervical spine surgery through the removal of the C3 is thought to give less damage to the muscles attached to the C2.
2. Purpose The aim of this study was to compare the prospective randomized comparison of these two surgical methods.
3. Hypothesis There is no difference in the cervical length and overall cervical angle between 1 month, 3 months, 6 months, and 12 months postoperatively between C3 laminectomy with C4-6 laminoplasty and C3-6 laminoplasty.

DETAILED DESCRIPTION:
Surgery is performed under general anesthesia as before, followed by posterior cervical incision. In one group, the cervical spine of the C3 is removed using a drill and punch and C4-6 laminoplasty will be performed. In the other group, C3-6 laminoiplasty will be performed. Postoperative suturing and subject management are the same as existing patient care policies. Follow-up is performed at 1 month, 3 months, 6 months, 12 months, and 1 year after surgery at the outpatient clinic and x-ray is taken at each outpatient follow-up. The degree of the neck pain is measured using NDI and VAS for each outpatient f/u.

ELIGIBILITY:
Inclusion Criteria:

* cervical stenosis

Exclusion Criteria:

* metastatic tumor
* fracture
* previous cervical spine surgery (posterior approach)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cervical stenosis who should undergo cervical laminoplasty
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
neck pain | 1 year
  Numerical rating pain score on neck, 0~10, 0 is no pain, 10 is maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Chun Kee Chung, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No